CLINICAL TRIAL: NCT07284056
Title: Prevention and Treatment of Early Postoperative Atelectasis Using The MetaNeb System in Patients Underwent Esophagectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2024847
Record Dates: First submitted 2025-12-02; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Atelectases, Postoperative Pulmonary
MeSH Terms: conditions — Pulmonary Atelectasis | interventions — Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Group (Sham Comparator)
  Interventions: Behavioral: Standard of care
- MetaNeb Group (Experimental)
  Interventions: Device: MetaNeb Therapy

INTERVENTIONS:
Device: MetaNeb Therapy — Patients in the MetaNeb group receive at least 4 sessions of MetaNeb therapy on postoperative day 1 (each session includes cycles of CPEP and CHFO modes totaling 10 minutes).
  Arms: MetaNeb Group
Behavioral: Standard of care — Standard postoperative care, including guidance on coughing and expectoration, turning and back percussion, and early mobilization (getting out of bed for physical activity).
  Arms: Standard Group

SUMMARY:
The goal of this clinical trial is to evaluate whether the MetaNeb® System can effectively prevent and treat early postoperative atelectasis in adult patients admitted to ICU after esophagectomy for esophageal cancer.

The main question it aims to answer is: can the MetaNeb® system significantly reduce the lung ultrasound score (LUSS) indicating atelectasis on postoperative days 1 and 2? Participants will be randomly assigned to either the standard treatment or MetaNeb group, undergo lung ultrasound and electrical impedance tomography (EIT) assessments on postoperative days 1 and 2, receive at least 4 sessions of MetaNeb therapy on postoperative day 1 if in the intervention group, be monitored for oxygenation indices, ICU stay duration, incidence of mechanical ventilation, need for bronchoscopic intervention, and adverse events like pneumothorax.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 85 years.
2. Patients who are scheduled for ICU admission after esophagectomy for esophageal cancer.

Exclusion Criteria:

1. Presence of an artificial airway at the time of ICU admission.
2. Planned ICU stay less than 24 hours.
3. Patients with contraindications to the use of the MetaNeb® System, or those unable to cooperate due to organic or psychiatric conditions.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 178 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference of lung ultrasound scores (LUSS) indicating atelectasis on postoperative day 1 and 2 | From postoperative day 1 to day 2

SECONDARY OUTCOMES:
The difference of dorsal ventilation region assessed by electrical impedance tomography (EIT) on postoperative day 1 and 2 | From postoperative day 1 to day 2
The difference of PaO2/FiO2 ratios on postoperative day 1 and 2 | From postoperative day 1 to day 2
The number of cases that underwent bronchoscopy intervention during ICU stay | From admission to ICU discharge
The number of cases that underwent high flow oxygen therapy or mechanical ventilation | From admission to ICU discharge
Length of ICU stay | From admission to ICU discharge
The number of cases that develop pneumothorax during intervention | From admission to the end of intervention at postoperative day 2

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
It might compromise the interests of MetNeb company and we still need to negotiate it further.